CLINICAL TRIAL: NCT02370862
Title: A Novel Application of Iontophoresis in the Transcutaneous Delivery of a Prokinetic Agent for the Promotion of Bowel Evacuation
Brief Title: Transdermal Administration of a Prokinetic Agent for Bowel Evacuation in Persons With SCI
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Mark Korsten, Chief of Gastroenterology, James J. Peters Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KOR-13-02
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Spinal Cord Injury; Neurogenic Bowel
Keywords: Spinal Cord Injury; Neurogenic Bowel; Bowel Evacuation; Gut Motility
MeSH Terms: conditions — Spinal Cord Injuries; Neurogenic Bowel | interventions — Neostigmine; Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bowel Evacuation Study with NEO and GLY (Experimental): The study design will consist of a screening visit to determine each individual's response to a previously established IV dose of NEO and GLY, followed by a dose titration study (two visits) of iontophoresed NEO and GLY. Study visits will be separated by no less than 2 days and no more than 14 days.
  Interventions: Drug: Neostigmine and Glycopyrrolate

INTERVENTIONS:
Drug: Neostigmine and Glycopyrrolate

SUMMARY:
Bowel care (BC) is a time-consuming and cumbersome activity of daily living for most individuals with SCI. Previous studies have reported that the average time to complete a BC routine is 45 minutes; 10-20% of SCI individuals report BC routines lasting for more than 1 hour. In past studies, the investigators have shown that a medication called neostigmine (NEO) combined with a medication called glycopyrrolate (GLY) can increase bowel activity and thus, promote bowel movement. The investigators have successfully used this medication with traditional and novel methods of colonoscopic preparations, and have shown that it improves the quality of these preparations. In this Phase I, proof of concept pilot study, the investigators propose to study the effectiveness of this medicine when it is delivered through the skin. In order to make delivery more efficient, the investigators will be using a technique called iontophoresis, which uses a mild electric current to drive the drug through the surface of the skin. The instrument includes an electrode containing the active agent (delivers charge) and an oppositely charged electrode (receives charge) which will be placed on the surface of the skin. The study design will consist of a screening visit to determine each individual's response to a previously established IV dose of NEO and GLY, followed by a dose titration study (two visits) of iontophoresed NEO and GLY. Study visits will be separated by no less than 2 days and no more than 14 days.

If this delivery method is shown to be effective, it may represent a way to vastly improve the clinical utility of this medication by allowing for needle-free self administration, and expanding the clinical indication to routine, at home bowel care.

DETAILED DESCRIPTION:
In this Phase I, proof of concept pilot study, we propose to study the safety and efficacy of transcutaneous neostigmine and glycopyrrolate facilitated by iontophoresis. The study design will consist of a screening visit to determine each individual's response to a previously established IV dose of NEO and GLY, followed by a dose titration study (two visits) of iontophoresed NEO and GLY. Study visits will be separated by no less than 2 days and no more than 14 days.

Screening Bowel Evacuation Study, Part 1: Visit 1 (30 Subjects with SCI):

A previously determined efficacious dose of IV neostigmine (0.03 mg/kg IV NEO) with glycopyrrolate (0.006 mg/kg GLY) will be administered during the first study visit to determine subject responsiveness to the known effective mode of administration. Irregardless of excess weight, the maximum dose of neostigmine and glycopyrrolate (NG) is limited to 10.0 mg and GLY to 2.0 mg. If the subject responds to the IV NEO, subsequent study visits to determine the effective dose of transcutaneous NEO and GLY will be performed. Subjects will be asked to arrive at the Spinal Cord Research Center at the James J. Peters Veteran Affairs Medical Center (JJP VAMC) (Room 7A-13) on the day of their scheduled study visits. Heart rate (continuous ecg), blood pressure, airway resistance (Impulse Oscillometry, IOS), signs and symptoms, and artificial bowel evacuation will be monitored throughout the study visit. Subjects will remain in this position until a bowel movement occurs, or for the next 60 minutes of the study. Subjects will be monitored for a minimum of 1.5 hours post drug, and until they reach ± 10% of their baseline heart rate (continuous 3 lead ECG) and airway caliber as measured by IOS.

Transcutaneous Bowel Evacuation Study, Part 2: Visits 2-3 (up to 25Subjects with SCI):

The same subjects who participated in Visit 1 who demonstrated a response to the IV NEO and GLY will participate in visits 2-3. Due to probable inter-subject variability of drug response to the doses of neostigmine being administered, subjects will receive increasing doses of iontophoresed neostigmine on separate days over 2 study visits to determine the most effective average dose. We will administer the transcutaneous NEO and GLY facilitated by iontophoresis. The dosages for Visits 2-3 are as follows: Visit 2: 0.05 mg/kg NEO and 0.01 mg/kg GLY, Visit 3: 0.07 mg/kg NEO and 0.14 mg/kg GLY. Irregardless of excess weight, the maximum dose of NG is limited to 10.0 mg and GLY to 2.0 mg. Heart rate (continuous ecg), blood pressure, airway resistance (Impulse Oscillometry, IOS) signs and symptoms, and artificial bowel evacuation will be monitored throughout the study visit as described in Table 1. Subjects will be asked to arrive at the Spinal Cord Research Center at the JJP VAMC (Room 7A-13) on the day of their scheduled study visits. Subjects will remain in this position until a bowel movement occurs, or for the next 90 minutes of the study. Subjects will be monitored for a minimum of 90 minutes post drug, and until they reach ± 10% of their baseline heart rate (continuous 3 lead ECG) and airway caliber as measured by IOS.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete or complete SCI,
* Tetraplegia or paraplegia,
* Excess time for bowel evacuation (> 60 minutes per bowel training session)

Exclusion Criteria:

* Previous adverse reaction or hypersensitivity to electrical stimulation,
* Known sensitivity to neostigmine or glycopyrrolate,
* Do not require additional bowel care or have "normal bowel function",
* Blockage Bowel or Bladder,
* Myocardial infarction in the past 6 months,
* Blood pressure of 160/100mmHg or higher with or without being on 3 or more different classes of anti-hypertensive medications
* Organ damage (heart & kidney damage) and/or transient ischemic attack (TIA)- cerebrovascular accident (CVA) as a result of hypertension
* Known past history of coronary artery disease or bradyarrythmia,
* Active respiratory disease,
* Known history of asthma during lifetime or recent (within 3 months) respiratory infections.
* Adrenal insufficiency,
* Pregnancy or potential for pregnancy,
* Lactating/nursing females,
* Slow heart rate (<45 bpm)
* Use of any antibiotic in the past 7 days,
* Use of medications known to affect the respiratory system,
* Use of medications known to alter airway caliber,
* Concurrent participation in other clinical trials (within 30 days).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Biological Responses to Study Drugs (quantified by the presence and strength of biological responses (changes in bowel sounds, heart rate and airway resistance and bowel movement occurrence) | 6 months
  We aim to determine the efficacy of transcutaneous (TC) neostigmine (NEO) with glycopyrrolate (GLY) delivered via iontophoresis in promoting bowel movement in persons with chronic SCI. This will be quantified by the presence and strength of biological responses (changes in bowel sounds, heart rate and airway resistance and bowel movement occurrence).

SECONDARY OUTCOMES:
Safety of Study Medication (quantified through monitoring of side effects during study visits and through patient self report as measured by the Treatment Satisfaction Questionnaire) | 6 Months
  We aim to determine the safety and tolerability of TC NEO and GLY in persons with SCI when used to promote bowel movement. This will be quantified through monitoring of side effects during study visits and through patient self report as measured by the Treatment Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Korsten, MD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States